CLINICAL TRIAL: NCT05391919
Title: Multimodal Correction of Post-stroke Motor and Cognitive Impairments With the Integrated Use of Innovative Digital Technologies, Biofeedback, Virtual Reality, a Neurointerface With Cardiovascular Risks Monitoring in an Outpatient Clinic
Brief Title: Multimodal Correction of Post-stroke Motor and Cognitive Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine (Other)
Collaborators: Moscow Government (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/17.03.2022
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Stroke Rehabilitation
Keywords: ischemic stroke rehabilitation; post-stroke dysfunction of the hand; cognitive disfunction; artificial intelligence; virtual reality; neurointerface; smart glove; biofeedback; cardiology risk control; upper limb medical rehabilitation; digital interactive technology

STUDY DESIGN:
Intervention Model Description: Open lable randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MT in early recovery period of IS (Experimental): Patients in early recovery period of IS receive a course of rehabilitation with multimodal correction using BFB-stabilometric training, cognitive-motor training in a virtual environment (VR), functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator "SensoRehab", if moderate paresis of the upper limb - the neurointerface "Exokist-3" with EEG registration.
  Interventions: Other: Multimodal technology (MT)
- MT in late recovery period of IS (Experimental): Patients in late recovery period of IS receive a course of rehabilitation with multimodal correction using BFB-stabilometric training, cognitive-motor training in a virtual environment (VR), functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator "SensoRehab", if moderate paresis of the upper limb - the neurointerface "Exokist-3" with EEG registration.
  Interventions: Other: Multimodal technology (MT)
- No MT Intervention: Conventional IS rehabilitation (Active Comparator): Patients in early and late recovery period of IS recieve conventional complex rehabilitation: kinesiotherapy, physiotherapy, occupational therapy.
  Interventions: Other: Conventional rehabilitation (CR)

INTERVENTIONS:
Other: Multimodal technology (MT) — Patients will receive a course of rehabilitation with multimodal correction using BOS-stabilometric training, cognitive-motor training with double and triple tasks once a day for the affected hand, virtual reality, functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator "SensoRehab", in moderate paresis of the upper limb, the neurointerface "Exokist-3" with EEG registration will be used. The program for IS patients includes 15 sessions with the MT: 15-30 minutes every method 2-3 times a week, 5-8 weeks.The total duration of one procedure is 2-3 hours.
  Arms: MT in early recovery period of IS; MT in late recovery period of IS
Other: Conventional rehabilitation (CR) — The patients will recieve Conventional rehabilitation technology (physiotherapy, kinesiotherapy, occupational therapy. The program for IS patients includes 15 sessions with the CR: 15-30 minutes every method 2-3 times a week, 5-8 weeks.The total duration of one procedure is 2-3 hours.
  Arms: No MT Intervention: Conventional IS rehabilitation

SUMMARY:
The aim of the study is the development and scientific substantiation of the effectiveness and safety of multimodal rehabilitation technology using innovative digital technologies, biofeedback (BFB), virtual reality (VR), neurointerface for the restoration of stato-locomotor disorders, neuromuscular control of upper limb movements and cognitive functions in patients with ischemic stroke (IS) in different recovery periods with rehabilitation risks control in outpatient clinic.

DETAILED DESCRIPTION:
The object of the study The study will include 90 patients (men and women) with the diagnosis of ischemic stroke (IS) in the early recovery (up to 6 months) and late recovery (6-12 months) periods with stato-locomotor disturbances, dysfunction (violation of neuromuscular movement control) of the upper limb (UL), mild or moderate cognitive impairment.

Patients will be randomly assigned to one of three experimental groups - 2 main groups in the early (30 patients) and in the late recovery period (30 patients) of IS and 1 comparison group (30 patients) in the early and late recovery periods of IS.

Each participant of the study will be assigned an ordinal number. Patients of the 1st and 2nd main groups are planned to undergo a rehabilitation course with multimodal correction, depending on the severity of functional and neuropsychological disturbances with the use of FBF-stabilometric training, cognitive-motor training with double and triple tasks in a virtual environment, functional individually programmed stimulation of antagonist muscles of the lower limb (FES), training of subject-manipulative activity for the restoration of fine hand movements on the glove simulator "SensoRehab"; when severe and moderate paresis of the upper limb, the neurointerface "Exokist-3" with EEG registration will be used.

The mode of application of multimodal correction technology: 15 procedures, 2-3 times a week, the duration of the course is 5-8 weeks. The total duration of one procedure is 2-3 hours a day.

Multimodal correction technology will not be included in the rehabilitation program of patients in the comparison group.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 45 to 70 years after a first-onset IS, early (1-6 months), late recovery (6-12 months) periods.
2. Supratentorial IS according to MRI of the brain.
3. The severity of UL paresis ranged from a score of 4 to 3 according to the Medical Research Council Scale (MRCS).20
4. Spasticity of 2 points or less by the Modified Ashworth Scale (MAS)
5. Cognitive function more than 20 points on the Montreal Cognitive Assessment (MoCA)
6. Affective disorders score less than 11 on the Hospital Anxiety and Depression Scale (HADS)
7. The patient's ability and willingness to comply with the requirements of this protocol.

Exclusion Criteria:

1. Concomitant neurological diseases causing decreased muscle strength or increased muscle tone in the UL (e.g., cerebral palsy, brain injury).
2. Clinically significant limitation of the passive movement amplitude in the joints of the investigated hand, pronounced contracture and deformities of the upper extremity.
3. Use of other DIT, BFB techniques to restore impaired UL function within 30 days prior to the patient Inclusion Visit.
4. Severe visual impairment, decreased visual acuity of less than 0.2 in the worst eye according to the Golovin-Sivtsev Table24.
5. Sensory aphasia, gross motor aphasia.
6. Recurrent stroke.
7. Epilepsy
8. Unstable angina and/or heart attack in previous month.
9. Uncontrolled arterial hypertension.
10. Somatic diseases in decompensation stage.
11. Thrombosis of deep and superficial veins of the lower extremities
12. The presence of left-handedness in the patient according to the Edinburgh manual asymmetry questionnaire
13. Alcohol abuse, medical marijuana use or soft drug abuse within the 12 months prior to the Inclusion Visit.
14. Any medical condition, including mental disease or epilepsy that could affect the interpretation of study results, the study procedures or patient safety.

15 Pregnancy. 16. Lactation.

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Scale (FMA-UE) dynamic | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  The FMA UE Scale comprises 33 items, each scored on a scale of0 to 2, where 0 = cannot perform, 1 = performs partially and2 = performs fully. It is free, requires only household items fortesting, and takes up to 30 minutes to administer. Changes in sections A-D of the FMA-UE Scale by 7 points or more are considered as efficacy.
Action Research Arm Test (ARAT) Scale dynamic | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  The Action Research Arm Test (ARAT) is a 19 item observational measures. Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally). Changes in the total ARAT Scale score by 4 points or more more are considered as efficacy.
Change from Baseline in 10 Metre Walk Test | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  The individual walks without assistance for 10 meters, with the time measured for the intermediate 6 meters to allow for acceleration and deceleration. The total time taken to ambulate 6 meters is recorded Timing starts when the toes pass the 2-meter mark Timing stops when the toes pass the 8-meter mark
Change from Baseline in Tinetti test | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  The Tinetti-test is used to assess the gait and balance, perception of balance and stability during activities of daily living.The Tinetti test has a gait score and a balance score. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the Tinetti test, the higher the risk of falling.
Changes in cognitive status | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  Assesment by the Montreal Cognitive Assessment scale (МоСА). MoCA is scored out of 30. A cut-off score of 26 signifies mild cognitive impairment.
Change from Baseline of Presence and severity of depression and anxiety | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  The Hospital Anxiety and Depression Scale (HADS). Changes in HADS anxiety and depression scores.The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.8-10 - points subclinically expressed anxiety / depression 11 points and above - clinically expressed anxiety / depression.
Restoration of CNS function | Baseline, day 15 of MT
  Concentration of human brain neurotrophic factor (BDNF) in the blood serum of patients by solid-phase enzyme immunoassay

SECONDARY OUTCOMES:
Percentage of correctly performed tasks | Baseline, day 7, day 15
  percentage of correctly performed tasks while training
change in the paresis degree ин the 6-point Medical Research Council Scale for assessing muscle strength: MRCS | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  The 6-point Medical Research Council Scale for assessing. The patient's effort is graded on a scale of 0-5. Grade 5: Muscle contracts normally against full resistance.Grade 0: No movement is observed. Grade 4 - light paresis. Grade 3 - moderate paresis. Grades 1-2 - severe paresis. The best result is 5, deterioration - a decrease in the indicator on the scale
Changes in spasticity severity | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  Modified Ashworth Scale: MAS (0 to 4 points). Scoring: 0 No increase in tone (the best point); 4 limb rigid in flexion or extension (the worse outcome)
Changes in level of impairment or dependence in daily life | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  Barthel Index.The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.Each item is rated in terms of whether the patient can perform the task independently, with some assistance, or is dependent on help based on observation (0=unable, 1=needs help, 2=independent). The final score is x 5 to get a number on a 100 point score. Proposed guidelines for interpreting Barthel scores are that scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency.
Changes of Life quality assessment | Baseline, day 7, day 15 of MT and 6 weeks after completing training
  European Quality of Life Questionnaire EuroQol EQ-5D-5L (version 1.0, 2011 in combination with the visual analogue scale). Health State: The respondent classifies his or her prevailing state of health by selecting one of three different levels of problem severity within each of five health domains. The levels are none, moderate and severe/extreme (coded 1 through 3, respectively), whilst the domains are mobility, capacity for self-care, conduct of usual activities, pain/discomfort and anxiety/depression, ordered as such.
  Evaluation: The respondent then evaluates his or her health using a visual analogue scale (VAS). This is a vertical, calibrated, line, bounded at 0 ("worst imaginable health state") and at 100 ("best imaginable health state"). Respondents indicate where they perceive their present state of health to lie, relative to these anchors.
Canges in Rehabilitation routing scale. | Baseline, day 15 of MT and 6 weeks after completing training
  The rehabilitation Routing Scale (SRM), developed by the Ministry of Health of Russia has six points:
  1. The absence of significant disorders of vital activity, despite the existing symptoms of the disease
  2. Slight restriction of vital activity
  3. Restriction of vital activity, moderate in its severity
  4. Pronounced restriction of vital activity
  5. Gross violation of vital processes
  6. Violation of vital activity of extreme severity An improvement is considered to be a decrease in the score on the scale.
Changes by international scale of functioning, disability and health (ISF) | Baseline, day 15 of MT and 6 weeks after completing training
  A generic qualifier scale can be used to record the extent of the problem for each identified impairment, activity limitation and participation restriction. Environmental factors can also be qualified as either barriers or facilitators. Improvement - reduction of the qualifier's score in the selected domain

OTHER OUTCOMES:
Number of participants with abnormal electrocardiogram (ECG) readings | Baseline, day 1-15 of MT
  Cases of ECG deviations during the MT session are taken into account (for example, ST segment changes, occurrence of arrhythmia, QT Interval)
Number of participants with abnormal electroencephalogram (EEG) readings | Baseline, day 15 of MT
  Cases of ECG deviations during the MT session are taken into account (paroxysmal activity)

CONTACTS AND LOCATIONS:
Overall Officials: Elena V Kostenko, PhD, D. Sс (Medicine), Study Director — Moscow scientific and practical center of medical rehabilitation, restorative and sports medicine of the Department of health of the city of Moscow, branch 7;
Locations (1):
- Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine, branch 7, Moscow, Russia